CLINICAL TRIAL: NCT01432873
Title: A Randomized Double Blinded Placebo Controlled Oral Selenium Therapy for the Prevention of Mucositis in Patients Undergoing High Dose Chemotherapy With Hematopoietic Stem Cell Transplantation
Brief Title: Oral Selenium Therapy for the Prevention of Mucositis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HORCSCT-9001
Record Dates: First submitted 2011-07-25; First posted 2011-09-13 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Mucositis; Hematopoietic Stem Cell Transplantation
Keywords: BMT; HSCT
MeSH Terms: conditions — Mucositis | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Oral selenium therapy arm
  Interventions: Drug: Oral selenium
- Placebo (Placebo Comparator): Oral placebo
  Interventions: Drug: Oral placebo

INTERVENTIONS:
Drug: Oral selenium — Drug: selenium tablet Oral selenium 1 Tab bid from day -6/-7 until discharge
  Arms: Experimental
Drug: Oral placebo — Drug: Placebo Oral placebo 1 Tab bid from day -6/-7 until discharge
  Arms: Placebo

SUMMARY:
Selenium as an antioxidant and anti-inflammatory agent could be effective in prevention of mucositis induced by chemotherapy and radiotherapy. Other agents such as vitamin E, Zinc sulfate, amifostine, beta carotene and benzidamine are indicated for prevention of mucositis and positive effects are seen. Our purpose in this double blinded randomized study is to evaluate the selenium effect on mucositis prevention in patient with acute myeloid leukemia (AML) & acute lymphoblastic leukemia (ALL) whose received Busulfan and/or Cyclophosphamide before Hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Patients with AML or ALL diagnosis, candidates for high dose chemotherapy with stem cell transplantation will be screened for enrollment in the study.

Patients will be randomized in two groups with balanced block randomization method. One group will receive selenium tablet twice per day and another group will receive placebo two times per day.Therapy will start on the morning before starting chemotherapy and will continue until the first of either discharge day or day +21.

Response assessment will include:

1. Mucositis assessment using WHO grading and OMAS scores- to be done from baseline and until day +21 or discharge day if before day +21.
2. Evaluation of selenium and glutathione peroxidase levels in the serum, - to be done at baseline, day +7 and day +14.
3. Collection of clinical outcome data regarding infectious complications including- presence and length of febrile neutropenia, use of antibacterial and antifungal medications

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML or ALL undergoing high dose chemotherapy with stem cell transplantation
* Adequate renal and hepatic function

Exclusion Criteria:

* Taking selenium supplement before admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The grade of oral mucositis after bone marrow transplantation | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  The effect of oral selenium on prevention of mucositis in patients undergoing bone marrow transplantation

SECONDARY OUTCOMES:
Evaluation of selenium concentration and glutathione peroxidase level in serum | up to 3 weeks
Total days of mucositis after BMT | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Molouk Hadjibabaie, Pharma D, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Iran

REFERENCES:
- [Derived] Jahangard-Rafsanjani Z, Gholami K, Hadjibabaie M, Shamshiri AR, Alimoghadam K, Sarayani A, Mojtahedzadeh M, Ostadali-Dehaghi M, Ghavamzadeh A. The efficacy of selenium in prevention of oral mucositis in patients undergoing hematopoietic SCT: a randomized clinical trial. Bone Marrow Transplant. 2013 Jun;48(6):832-6. doi: 10.1038/bmt.2012.250. Epub 2013 Jan 7. PMID 23292233